CLINICAL TRIAL: NCT00720239
Title: Safety and Wound Healing Efficacy of the TalidermR Wound Dressing a Poly-N-acetyl Glucosamine-derived Membrane Material in Humans With Venous Stasis Ulcers: a Pilot Study.
Brief Title: Taliderm Dressing for Venous Ulcers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Teresa Kelechi, Professor, Medical University of South Carolina
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86606
Record Dates: First submitted 2008-02-07; First posted 2008-07-22 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Venous Stasis Ulcers; Venous Insufficiency
MeSH Terms: conditions — Varicose Ulcer; Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0 (No Intervention)
- 1 (Experimental): Experimental Group 1 (n = 10) will receive TalidermR to the wound once during the treatment phase.
  Interventions: Other: Taliderm wound healing dressing
- 2 (Experimental): Experimental Group 2 (n = 10) will receive TalidermR to the wound every other week during the treatment phase.
  Interventions: Other: Taliderm wound healing dressing
- 3 (Experimental): Experimental Group 3 (n = 10) will receive TalidermR to the wound every three weeks during the treatment phase.
  Interventions: Other: Taliderm wound healing dressing

INTERVENTIONS:
Other: Taliderm wound healing dressing — Taliderm wound healing dressing will be applied to the wound site as follows depending on assignment to group:
  Control group receives no intervention. Experimental Group 1 (n = 10) will receive TalidermR only one time at the beginning of the treatment phase.
  Experimental Group 2 (n = 10) will receive TalidermR to the wound every other week during the treatment phase.
  Experimental Group 3 (n = 10) will receive TalidermR to the wound every three weeks during the treatment phase.
  Arms: 1; 2; 3

SUMMARY:
The study will test a new wound healing dressing called Taliderm® on leg ulcers caused by chronic venous insufficiency (CVI). Some people with CVI have poor vein circulation that causes ulcers to develop on the lower legs. This new dressing is hoped to help the ulcers heal more quickly. The study hypothesis is to determine whether the TalidermR Wound Dressing, a poly-N-acetyl glucosamine (pGlcNAc) derived membrane material expedites wound healing in humans with venous stasis ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥45 years of age
* Diagnosis venous partial thickness ulcer diagnosed within the past
* 4 weeks without recent enzymatic, autolytic or chemical treatment
* Viable and clean wound bed with granulation tissue and ≥ 90% free of necrotic debris
* Wound measures between 5 and 20 cm2
* Extends through epidermis and into the dermis

Exclusion Criteria:

* Full thickness ulcers extending beyond the dermis
* Current wound, skin, or systemic infection
* Wound bed ≤90% free of necrotic debris
* Recent treatment with enzymatic, autolytic or chemical agents
* History or collagen vascular disease, severe arterial disease, organ transplant, Charcot, sickle cell
* Insufficient blood supply to ulcer (ankle-brachial index <.8 or >1.3)
* History of radiation therapy to the site
* Cellulitis/osteomyelitis/avascular ulcer bed
* Currently receiving hemodialysis
* Pregnancy
* Currently receiving treatment with another investigational drug or device or within the past 30 days
* Unable to comply with the study protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-02; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
wound healing | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Teresa J Kelechi, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Roper St. Francis Hospitals, Charleston, South Carolina, United States